CLINICAL TRIAL: NCT06548191
Title: TREAD: Time Restricted Eating Intervention for Alzheimer's Disease
Acronym: TREAD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Paula Desplats, Associate Professor of Neuroscience, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RD10061932; R61AG085253 (NIH)
Record Dates: First submitted 2024-07-20; First posted 2024-08-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Alzheimer's Disease
Keywords: Time-Restricted Eating; Intermittent Fasting; Prolonged Nightly Fasting; Mild Cognitive Impairment; Alzheimer Disease; Circadian Rhythms; Cognition; Neuropathology
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: TREAD will enroll 40 older adults (60+ years) with cognitive impairment and clinically diagnosed with Mild Cognitive Impairment (MCI) or early to moderate AD; and 20 cognitively normal subjects (18+ years). The investigators will recruit individual participants with a diagnosis of MCI/AD (n=20 subjects) and 20 dyads of participants (n=40 subjects) composed of an MCI/AD patient and a cognitively normal living partner. This design is necessary to evaluate how feasible and burdensome is to follow a time-restricted eating pattern for individuals with cognitive impairment. Individual and dyad participants will be randomized in equal ratios to the complete prolonged nightly fasting intervention (14 h fast with no energy intake after 8 pm for 6 months) or to a delayed-start prolonged nightly fasting intervention (3 initial months of unrestricted eating patterns followed by 3 months of 14 h fast with no energy intake after 8 pm) using a random permuted-block design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding disease condition and arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed-Start Intervention (Active Comparator): Participants will continue their regular eating schedule (nightly fasting for less than 12 h) during the first 3 months and start time-restricted eating intervention ( 14 h of nightly fasting) for the next 3 months.
  Interventions: Behavioral: Time-restricted eating
- Intervention (Active Comparator): Participants will follow the time-restricted regimen (14 h of nightly fasting) for 6 months.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Fasting (abstinence from calorie-containing food or drink) during 14 h at night, with no caloric consumption after 8 pm to align with circadian rhythms
  Other Names: Prolonged Nightly Fasting

SUMMARY:
The goal of this clinical trial is to learn if restricting the time of eating to allow for prolonged fasting at night may reduce sleep disturbances, cognitive decay, and pathology in patients diagnosed with Mild Cognitive Impairment (MCI) or early to moderate Alzheimer's disease (AD). It will also learn about the feasibility of practicing 14 h of nightly fasting in this group of older adults. The main questions it aims to answer are:

* Does prolonged nightly fasting of 14 h can reduce markers of AD pathology and aging and reduce cognitive and sleep alterations in MCI and AD patients?
* Can patients with MCI and early /moderate AD sustain time-restricted eating for 3 to 6 months? Researchers will compare participants who fast for 14 h per night during 3 months to those who fast for less than 12 h/night. Researchers will also compare participants that fast for 3 months to those who fast during 6 months, to determine the effective duration of the intervention. Finally, researchers will evaluate whether following the time-restricted eating diet alongside a partner actively following the same diet, will increase adherence to the protocol compared to subjects that fast alone.

Participants will:

* Fast for 14 h a night (stop eating at 8 pm and start eating the following morning at 10 am) for 3 or 6 months
* Visit the clinic three times (at the beginning of the study, 6 and 12 months later)
* Provide blood samples and take a cognitive test during clinic visits
* Keep a diary (or use an app on a smart phone) to record time of eating
* Wear an activity tracker watch

DETAILED DESCRIPTION:
Study Description: Our overarching hypothesis is that circadian alignment of food intake and biological clocks can reduce pathology and improve cognitive function in Alzheimer's disease (AD) patients. The rationale for this proposal is that the prolonged nightly fasting form of Time-restricted eating (TRE) aligns food intake with the daytime "wake phase" of the biological clock, optimizing nutrient processing, and may modulate disease trajectory in AD. This Pilot study will test the feasibility and safety of TRE, consisting of 14 hours of night fasting for 3 or 6 months, in patients along the AD continuum and will explore the outcomes of this intervention on markers of aging and AD pathology. Results from this study will provide a strong scientific justification and will optimize the methods for a larger trial to determine the clinical efficacy of TRE to mitigate disease progression in AD and related dementias.

Objectives:

Primary Objective: Test the feasibility of a TRE intervention (TREAD) among patients with Mild Cognitive Impairment (MCI) or AD.

Secondary Objectives: Explore the effects of TRE on metabolic and pathological markers in MCI/AD patients.

Endpoints:

Primary Endpoint: Feasibility, safety, cognition, and metabolic indicators. Secondary Endpoints: Biomarkers of AD pathology, sleep and activity, and markers of epigenetic aging.

Study Population:

Adult subjects (female and males, ≥60 years old) with normal cognition or with a clinical diagnosis of MCI/AD (meeting research consensus criteria for probable MCI or dementia due to AD).

Phase: Early phase 1

Description of Sites/Facilities Enrolling Participants:

Shiley-Marcos Alzheimer's disease Research Center (SMARDC) at the University of California San Diego (UCSD) La Jolla campus.

Description of Study Intervention: The investigators will enroll older-adult participants (>60 years old) clinically diagnosed with MCI or early to moderate AD (n=20 subjects) and 20 dyads of participants (n=40 subjects) composed of an MCI/AD patient and a cognitively normal living partner (> 18 years old ); for a total enrollment of 60 subjects. All participants must have a baseline nightly fasting of <12 h. Individual participants and dyads will be randomized into the Intervention group (INT) or the Delayed Start Intervention group (DS-INT). The intervention will involve prolonged nightly fasting of 14 hours (TRE). The INT group will follow the TRE regimen for 12 months. The DS-INT group will practice their regular eating pattern for 3 months (nightly fasting <12 h) followed by 3 months of TRE. All participants will have study visits, outcome assessments, and biospecimen collections at baseline, 3, and 6 months.

Study Duration: Two years Participant Duration: 6 months

ELIGIBILITY:
Provision of signed and dated informed consent form. Stated willingness to comply with all study procedures and availability for the duration of the study.

Inclusion criteria

1. Persons, aged ≥60 years
2. In good general health as evidenced by medical history or diagnosed with clinical diagnosis of MCI/AD: meeting research consensus criteria for probable MCI or dementia due to AD, requiring positive amyloid biomarkers in brain or cerebrospinal fluid (CSF) obtained at their regular point of care or study referral no longer than 3 months prior to screening.
3. Ability and willingness to complete cognitive evaluations, blood draw, actigraphy monitoring and to record fasting times daily.
4. Daily night fasting <12h at baseline. Ability and willingness to follow an eating protocol of prolonged night fasting for 14 h
5. For cognitively normal living partners in the dyads group, scores >26 in the Montreal Cognitive Assessment (MoCA) test administered at screening.

Exclusion Criteria:

1. Clinical diagnosis with a neurodegenerative condition other than MCI/AD.
2. Presenting cognitive impairment not due to AD.
3. Clinical diagnoses of diabetes.
4. Actively using insulin in the past 6 months.
5. Started a new medication (or changed doses) indicated for the treatment of MCI/AD in the last three months prior to enrollment.
6. Currently taking any medication known to affect appetite, inlcuding but not limited to GLP-1 agonists.
7. Any history of disordered eating, including difficulty swallowing and refusal to eat.
8. Currently engaged in shift work.
9. In treatment with another investigational drug.
10. Body Mass Index (BMI) <20. or >35

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: assessed by computing the number of nights achieving the goal fasting time of 14 h. | 3 and 6 months
  Test the feasibility of a Time-restricted eating intervention in patients with MCI or AD by quantification the number of days during the intervention period when the particpants reached the goal intervention fasting time of 14 h, b) increased fasting of >12 h and <14 h.

SECONDARY OUTCOMES:
Effects of TRE on activity rhythms measured as steps/day using an accelerometer | baseline, 3 and 6 months
  The investigators will measure the participants' 24-hour activity rhythms using an actigraph unit. The investigators will calculate interday stability and intraday variability of activity rhythms, which have been reported as sensitive in studies on aging and AD cohorts. Interday stability will indicate the stability of rhythms across several days. Intraday variability will indicate the fragmentation of rhythms.
Effects of TRE on skin temperature rhythms measured in F using a smart sensor. | baseline, 3 and 6 months
  The investigators will measure the participants' 24-hour temperature rhythms using a smart sensor. The investigators will calculate interday stability and intraday variability of skin temperature as a circadian output.
Effects of TRE on sleep quantity (as hours/night) using a smart sensor. | Baseline, 3 and 6 months
  The investigators will determine changes in sleep duration during the study as recorded by a smart sensor and accessed via the Fitabase.
Effects of TRE on sleep quality (determined by a sleep score) using a smart sensor. | baseline, 3 and 6 months
  The investigators will determine whether the overall sleep efficiency changes based on the sleep score calculated based on metrics collected with the accelerometer watch. The overall sleep score is a sum of the individual scores in sleep duration, sleep quality, and restoration, with a maximum of 100. Sleep score tiers are: Excellent: 90-100; Good: 80-89; Fair: 60-79; Poor: Less than 60.
Explore the effects of TRE on pathology in MCI/AD patients | baseline, 3 and 6 months
  Evaluate levels of amyloid Beta (AB)40, AB42, phospho-Tau181, Neurofilament light chain protein, and markers of neuroinflammation in plasma
Explore the effects of TRE on markers of epigenetic aging by profiling DNA methylation in blood samples. | baseline, 3 and 6 months
  The investigators will profile genome-wide DNA methylation in whole blood using the Infinium Methylation EPIC v2.0 array (Illumina) to determine whether prolonged fasting modulates epigenetic aging rates. A beneficial effect will result in no changes to the subjects' biological aging rate or a deacceleration of aging.
Explore the effects of TRE on fasting blood glucose (mg/mL) | baseline, 3 and 6 months
  The investigators will measure glucose levels in the blood at the end of fasting during the clinical visits to evaluate whether prolonged fasting reduces fasting glucose as an indicator of metabolic health.
Evaluation of neurocognitive changes using the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog). | baseline and 6 months
  The investigators will utilize the ADAS-Cog test to investigate whether TRE reduces cognitive decline in MCI and AD patients, expressed as the average score changes between visits. The ADAS-Cog is a brief neuropsychological assessment tool used to determine the severity of cognitive symptoms of dementia, widely used in clinical trials assessing antidementia treatments. The ADAS-Cog scores range from 0 to 70, with higher scores indicating poorer performance. It consists of 11 tasks, including Word Recall, Naming Objects and Fingers, Following Commands, Constructional Praxis, Ideational Praxis, Orientation, Word Recognition, Remembering Test Directions, Spoken Language, Comprehension, and Word-Finding Difficulty.
Evaluation of changes in self-reported sleep quality as determined by the Pittsburgh Sleep Quality Index (PSQI). | baseline, 3 and 6 months
  The investigators will utilize the PSQI to investigate whether TRE improves self-reported sleep quality. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the worst dysfunction. The global PSQI score ranges from 0 to 21 and is obtained by adding the scores of the seven components of the test. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Desplats, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Shiley Marcos Alzheimer's Disease Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared